CLINICAL TRIAL: NCT03603223
Title: A Phase II Open Label, Single Arm Study to Evaluate the Efficacy of Pembrolizumab for Leukoplakia
Brief Title: Pembrolizumab in Treating Participants With Leukoplakia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-001548; NCI-2018-01227 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pembrolizumab Leukoplakia; 16-001548 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2018-06-19; First posted 2018-07-27 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Erythroleukoplakia; Leukoplakia; Verrucous Oral Leukoplakia
MeSH Terms: conditions — Leukoplakia | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Participants receive pembrolizumab IV over 30 minutes on day 1. Courses repeat every 3 weeks for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II pilot trial studies how well pembrolizumab works in treating leukoplakia. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Clinical response rate at 6 months? percent of patients with complete response and partial response at 6 months.

SECONDARY OBJECTIVES:

I. Histologic response rate at 6 months. II. Change in clinical impression based on photographs of the lesion. III. Clinical response rate at 9 months and 12 months. IV. Toxicity.

EXPLORATORY OBJECTIVES:

I. PD-L1 expression in leukoplakia lesions and biomarker analysis.

OUTLINE:

Participants receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Courses repeat every 3 weeks for 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30 days and every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Subjects must have leukoplakia, erythroleukoplakia or proliferative verrucous leukoplakia (PVL) with lesions measurable in 2 dimensions, not amenable to surgical resection or radiation or who have refused surgery or radiation. Patients must have at least 1 lesion that can be followed on treatment. (Patients who have undergone complete excision of lesions and are clinically without evidence of disease will not be eligible for study.)
* Evidence of moderate or severe dysplasia or carcinoma in situ.
* Baseline biopsy specimen available for biomarker analysis or willingness to undergo fresh baseline biopsy.
* Willingness to consent to photographs of lesions.
* Willingness to undergo biopsy at 6 months.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale.
* Absolute neutrophil count (ANC) >= 1,500 /mcL within 10 days of treatment initiation.
* Platelets >= 100,000/mcL within 10 days of treatment initiation.
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment).
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (CrCl) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN within 10 days of treatment initiation. (Glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl).

  * Creatinine clearance should be calculated per institutional standard.
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN within 10 days of treatment initiation.
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamate pyruvate transaminase (SGPT) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases within 10 days of treatment initiation.
* Albumin >= 2.5 mg/dL within 10 days of treatment initiation.
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants. (Within 10 days of treatment initiation.)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants. (Within 10 days of treatment initiation.)
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 10 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Patients with leukoplakia, erythroleukoplakia or PVL who have only mild dysplasia or hyperplasia are excluded.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy > prednisone 10 mg daily or equivalent, or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus tuberculosis).
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject?s participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Has known active hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive) or hepatitis C virus (e.g., HCV ribonucleic acid [RNA] [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-05-03 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | At 6 months
  If there is a signal of efficacy based on this analysis, further exploratory analyses using Cox-proportional hazards regression, will be performed to identify variables which correlate to improved 6-month clinical response rate will be performed. Variables will include demographics, age, gender, pack-years smoking history, size of the lesions, prior history of leukoplakia or erythroleukoplakia, and human papillomavirus (HPV) status. While the study is not powered to detect a statistically difference between these groups, such an analysis may help identify a population more likely to benefit from treatment.

SECONDARY OUTCOMES:
Clinical response rate | At 9 and 12 months
  Response rate data will be reported in tabular form.

OTHER OUTCOMES:
PD-L1 positivity | Up to 2 years
  lesions will be stained to determine % PDL1 positivity
Correlation of response with PD-L1 positivity | Up to 2 years
  PDL1 positivity of the lesions will be correlated to response to pembrolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Wong, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (3):
- United States (3):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California